CLINICAL TRIAL: NCT03395327
Title: Pilot Study Describing the Early Evolution of the Sexual Function of Patients Receiving Adjuvant Hormone Therapy for Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CHD049-17
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: quality of life questionnaire — QLQ-C30 and BR23 (Quality of Life Questionnaire and Breast 23) Questionnaire FSFI (Female Sexual Function Index)

SUMMARY:
The 2014-2019 cancer plan emphasizes the need to "reduce the impact of cancer on personal life".

The impact of cancer on sexuality is multifactorial: fatigue, anxiety, impaired body image, chemotherapy treatment.

None of these studies specifically assessed the early impact on the quality of sexual life of patients.

The purpose of this study is to describe to describe the early evolution of the quality of sexual life of patients receiving adjuvant hormone therapy for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Female gender
* Histologically proven non-metastatic breast cancer
* Indication of adjuvant hormone therapy
* Patient able to understand a newsletter and to agree to participate

Exclusion Criteria:

* Age under 18 years
* Pregnant woman
* Adjuvant chemotherapy
* Patient followed for heavy psychiatric pathology (requiring guardianship or trusteeship)
* Persons protected or deprived of their liberty
* Male

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients managed for localized hormone-sensitive breast cancer but not receiving adjuvant chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2020-02-19 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
score FSFI (Female Sexual Function Index) | 3 month after adjuvant hormone therapy

CONTACTS AND LOCATIONS:
Locations (1):
- CHD Vendée, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No